CLINICAL TRIAL: NCT04148820
Title: One Versus Twice Daily Administration of Multiple Cardiovascular Agents in Patients With Ischemic Heart Disease: An Open Label, Randomized, Multicenter Study
Brief Title: One Versus Twice Daily Administration of Multiple Cardiovascular Agents in Patients With Ischemic Heart Disease
Acronym: ONCE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/D/789
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Ischemic Heart Disease
Keywords: coronary artery disease
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease | interventions — Aspirin; Atorvastatin; Perindopril

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Once daily drug administration (Experimental): Patients will be given cardiovascular drugs once daily
  Interventions: Drug: Aspirin, Atorvastatin, Perindopril
- Twice daily drug administration (Experimental): Patients will be given cardiovascular drugs twice daily
  Interventions: Drug: Aspirin, Atorvastatin, Perindopril

INTERVENTIONS:
Drug: Aspirin, Atorvastatin, Perindopril — Cardiovascular drugs will be administered all together every day at the same time

SUMMARY:
Patients with ischemic heart disease are often treated with multiple cardiovascular agents, including aspirin, statins, ezetimibe, Angiotensin Converting Enzyme (ACE) inhibitors or beta-blockers.

Uncertainty about the optimal timing and clinical implications of administration of cardiovascular drugs still persists.

The investigators will perform a pilot randomized trial to evaluate the efficacy and safety of a one daily administration of multiple drugs vs. twice daily administration.

DETAILED DESCRIPTION:
Patients with ischemic heart disease are often treated with multiple cardiovascular agents, including aspirin, statins, ezetimibe, Angiotensin Converting Enzyme (ACE) inhibitors or beta blockers.

These drugs are usually given at different timetables. Recent investigations, however, have demonstrated that adherence to medical treatment is significantly greater if a one daily strategy is adopted.

Uncertainty about the optimal timing and clinical implications of administration of cardiovascular drugs still persists.

The investigators will perform a pilot randomized trial to evaluate the efficacy and safety of a one daily administration of multiple drugs vs. twice daily administration.

ELIGIBILITY:
Inclusion Criteria:

Ischemic heart disease, willing to participate, compliance to medical therapy

Exclusion Criteria:

Patients with acute coronary syndrome; pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Outcome Event (MACE) | Up to 1 year
  The time to final occurrence of cardiovascular death, non-fatal myocardial infarction, ischemic stroke or ischemia-driven revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Marazzi, Study Director — San Raffaele Pisana
Locations (2):
- Italy (2):
  - San Raffaele Pisana, Rome
  - Sapienza University, Rome

IPD SHARING:
Plan to Share IPD: No